CLINICAL TRIAL: NCT00211510
Title: Use of the Paradigm 722 System to Improve Glycemic Control in Adult and Adolescent Subjects With Type 1 Diabetes: A Multi-center, Randomized Controlled Trial
Brief Title: Use of the Paradigm 722 System to Improve Glycemic Control in Adult and Adolescent Subjects With Type 1 Diabetes
Acronym: STAR1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP 178/Z25/A2
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Results first posted 2011-04-29 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes; Continuous Glucose Monitoring; Glycemic Control
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Paradigm 722 sensor augmented pump (Experimental): subjects will use the Paradigm 722 sensor augmented pump for infusion of insulin and continuous glucose monitoring
  Interventions: Device: Paradigm 722 sensor augmented pump
- Paradigm 715 insulin pump (Active Comparator): subjects will use the Paradigm 715 insulin pump which does not include sensor augmentation for infusion of insulin
  Interventions: Device: Paradigm 715 insulin pump

INTERVENTIONS:
Device: Paradigm 722 sensor augmented pump — Subjects use the Paradigm 722 sensor augmented pump
  Other Names: 722 pump
  Arms: Paradigm 722 sensor augmented pump
Device: Paradigm 715 insulin pump — Subjects use the Paradigm 715 insulin pump
  Other Names: 715 pump
  Arms: Paradigm 715 insulin pump

SUMMARY:
The purpose of this study is to determine whether Type 1 Diabetic subjects using the Paradigm 722 System, which is a glucose sensor-augmented insulin pump, can improve glycemic control when compared to subjects using the Paradigm 715 insulin pump only.

DETAILED DESCRIPTION:
Glycemic control remains a significant challenge for both adult and adolescent Type 1 diabetics. Continuous Glucose Monitoring (CGMS) is currently used by clinicians to record continuous, retrospective glucose measurements which aid in identification of glycemic excursion patterns. This data is then used to make therapy change recommendations for the future. The Paradigm 722 System transmits real-time glucose measurements to the insulin pump every 5 minutes, allowing users to view their current glucose values, as well as to review glycemic excursions and trends over a 24-hour period. This System will alert users to high and low glucose levels, and will allow subjects and their clinicians to treat to a therapeutic target HbA1c under monitored conditions.

Subjects wearing the Paradigm 722 System will be compared to subjects wearing the Paradigm 715 Insulin Pump over a 6 month period to evaluate changes in glycemic control (HbA1c).

ELIGIBILITY:
Inclusion Criteria:

* Age 12 - 80 years
* Type 1 Diabetes Mellitus diagnosed at least 1 year ago
* Using insulin infusion pump for past 6 months minimum
* Performing minimum 4 blood glucose tests per day
* Agree to treat to A1c targets
* Read and understand English

Exclusion Criteria:

* Pregnant or planning pregnancy
* History of unresolved tape allergy or skin conditions

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2005-06; Primary Completion 2006-08 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Lee, MD, Study Director — Medtronic
Locations (7):
- United States (7):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Stanford University, Stanford, California
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Joslin Diabetes Center, Boston, Massachusetts
  - The Endocrine Group, Albany, New York
  - Diabetes and Glandular Diabetes Research Associates, San Antonio, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Paradigm 722 Sensor Augmented Pump: subjects will use the Paradigm 722 sensor augmented pump for insulin infusion and continuous glucose monitoring
- Paradigm 715 Insulin Pump: subjects with use the Paradigm 715 insulin pump for insulin infusion
Period: Overall Study
Arm/Group | Paradigm 722 Sensor Augmented Pump | Paradigm 715 Insulin Pump
Started | 72 | 74
Completed | 66 | 72
Not Completed | 6 | 2
Not completed — Physician Decision | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Paradigm 715 Insulin Pump: subjects will use the Paradigm 715 insulin pump for insulin infusion
- Total: Total of all reporting groups
Arm/Group | Paradigm 722 Sensor Augmented Pump | Paradigm 715 Insulin Pump | Total
Number analyzed (Participants) | 72 | 74 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 23 | 43
  Between 18 and 65 years | 52 | 51 | 103
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (14.6) | 32.9 (16.3) | 32.4 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 46 | 84
  Male | 34 | 28 | 62
Region of Enrollment [Number; unit: participants]
  United States | 72 | 74 | 146

OUTCOME MEASURES:

1. Primary Outcome: Change in A1c From Baseline to 26 Weeks
Description: Change is defined as A1c at Week 26 minus A1c at Baseline in each study arm. The difference between the change in each group will then be analyzed. A1c measure is defined as the percent of glycated hemoglobin using one standardized assay for all subjects.
Time Frame: Baseline and 26 weeks
Measure: Mean (Standard Deviation); unit: Percent glycated hemoglobin
Arm/Group | Paradigm 722 Sensor Augmented Pump | Paradigm 715 Insulin Pump
Number analyzed (Participants) | 72 | 74
Percent glycated hemoglobin | -0.72 (0.69) | -0.58 (0.73)

2. Secondary Outcome: Difference in Frequency of Severe Hypoglycemia From Baseline to Week 26
Description: Severe Hypoglycemia as defined by hypoglycemic events requiring the assistance of another person to actively administer carbohydrates, glucagon or other resuscitative actions, as reported by subject. The frequency evaluates the total number of events. This will be analyzed and compared between the two study arms from baseline to week 26.
Time Frame: Baseline and 26 weeks
Measure: Number; unit: hypoglycemic events
Groups:
- Paradigm 715 Insulin Pump: subjects will use the Paradigm 715 pump for insulin infusion
Arm/Group | Paradigm 722 Sensor Augmented Pump | Paradigm 715 Insulin Pump
Number analyzed (Participants) | 72 | 74
hypoglycemic events | 11 | 3

3. Secondary Outcome: Changes in Hypoglycemia Area Under the Curve (AUC) From Baseline to Week 26
Description: Hypoglycemia is defined as a recorded blood glucose event <70mg/dL. The amount of time spent below this parameter will be analyzed and compared between groups from Baseline to Week 26
Time Frame: Baseline and 26 weeks
Measure: Mean (Standard Deviation); unit: mmol/dl*min
Arm/Group | Paradigm 722 Sensor Augmented Pump | Paradigm 715 Insulin Pump
Number analyzed (Participants) | 72 | 74
mmol/dl*min | -0.07 (0.581) | 0.281 (1.023)

4. Secondary Outcome: Changes in Hyperglycemia Area Under the Curve (AUC) From Baseline to Week 26
Description: Hyperglycemia is defined as a recorded blood glucose event > 180 mg/dL. The amount of time spent above this parameter will be analyzed and compared between groups from Baseline to Week 26
Time Frame: Baseline and 26 weeks
Measure: Mean (Standard Deviation); unit: mmol/dl*min
Groups:
- Paradigm 722 Sensor Augmented Pump: subjects with use the Paradigm 722 sensor augmented pump for insulin infusion and continuous glucose monitoring
Arm/Group | Paradigm 722 Sensor Augmented Pump | Paradigm 715 Insulin Pump
Number analyzed (Participants) | 72 | 74
mmol/dl*min | -10.2 (18.6) | -9.2 (16.2)

5. Secondary Outcome: Glucose Sensor Accuracy as Measured in the 722 Group
Description: Percent comparative sensor glucose reading to blood glucose meter in agreement within +/- 20% (Clark Error Grid zone A + zone B).
Time Frame: Baseline and 26 weeks
Measure: Number; unit: percent of agreement
Arm/Group | Paradigm 722 Sensor Augmented Pump | Paradigm 715 Insulin Pump
Number analyzed (Participants) | 72 | 74
percent of agreement | 95.9 | NA — Subjects in the Paradigm 715 arm did not wear the sensor and so no sensor accuracy could be tested.

6. Secondary Outcome: Problem Areas in Diabetes (PAID) Questionnaire Assessed and Compared Between Groups
Description: Questionnaire evaluating subjects'potential fear of hypoglycemia events. Change assessed at Baseline and Week 26 and compared between groups. Likert scale scored with 4 being the worst and 0 being no problem.
Time Frame: Baseline and 26 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Paradigm 722 Sensor Augmented Pump: subjects will use the Paradigm 711 sensor augmented pump for insulin infusion and continuous glucose monitoring
Arm/Group | Paradigm 722 Sensor Augmented Pump | Paradigm 715 Insulin Pump
Number analyzed (Participants) | 72 | 74
Scores on a scale | -0.07 (0.64) | -0.22 (0.66)

ADVERSE EVENTS:
Time Frame: Severe adverse event data and adverse device effects were collected for the six month study phase and six month continuation phase that followed.
Description: Some hypoglycemia events were self reported and unable to be independently evaluated or verified by the PI, while others had supporting clinical data. Those with supporting data are reported as Systematic, while the self reported events are reported as Non-systematic.
Arm/Group | Paradigm 722 Sensor Augmented Pump | Paradigm 715 Insulin Pump
Serious Adverse Events (participants affected / at risk) | 14/72 | 8/74
Other Adverse Events (participants affected / at risk) | 25/72 | 7/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paradigm 722 Sensor Augmented Pump (N=72) | Paradigm 715 Insulin Pump (N=74)
Severe Hypoglycemia (Endocrine disorders) | 10 (15) | 3 (6)
Diabetic Ketoacidosis (Endocrine disorders) | 3 (3) | 1 (1)
Skin abscess (Infections and infestations) | 1 (2) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Puncture wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paradigm 722 Sensor Augmented Pump (N=72) | Paradigm 715 Insulin Pump (N=74)
Haemorrhage (Vascular disorders) | 5 (8) | 3 (7) — Bleeding at sensor insertion site
Skin Irritation (Skin and subcutaneous tissue disorders) | 13 (15) | 4 (5)
Infection (Infections and infestations) | 4 (4) | 0 (0)
Pain (General disorders) | 3 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less